CLINICAL TRIAL: NCT07121218
Title: Assessment of Physical Fitness Level and Its Relationship With Pulmonary Functions in Patients With Bronchiectasis
Brief Title: Determination of Physical Fitness Level in Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: Melis Usul (Other)
Responsible Party: Sponsor-Investigator, Melis Usul, **Specialist Physiotherapist**, Istanbul Kent University
Organization: Istanbul Kent University (Other)
Other Study IDs: E-10420511-051-43479
Record Dates: First submitted 2025-08-03; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Patients With Bronchiectasis
Keywords: bronchiectasis; Physical Fitness
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with bronchiectasis
- Healthy individuals

SUMMARY:
The aim of this study is to assess the physical fitness level of children with bronchiectasis. To determine your physical fitness level, we will conduct some game-like tests. These are completely fun and enjoyable tests (such as running or a sit-to-stand test). Additionally, we will ask you some questions. These questions will help us get to know you better and understand how much you enjoy exercise. To measure your growth level, we will weigh you using a scale. We will also assess your muscle strength using a special device. All these tests will help us understand how much your condition affects you.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 18 years diagnosed with bronchiectasis
* Able to walk, cooperative, and clinically stable
* Children who can read and understand Turkish

Exclusion Criteria:

* History of lung transplantation
* Having experienced an acute exacerbation and/or hospitalization within the past month
* Having a musculoskeletal pathology that may affect mobility
* Presence of serious cardiac or neurological disease

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 7 to 18 years diagnosed with bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
FitnessGram Physical Activity Test Battery | Baseline (day of enrollment) assessment
Pulmonary function test | Baseline (day of enrollment) assessment
Peripheral Muscle Strength | Baseline (day of enrollment) assessment

SECONDARY OUTCOMES:
Physical Activity Level | Baseline (day of enrollment) assessment
  Physical activity level will be assessed using the Children's Physical Activity Questionnaire (CPAQ) developed by Kowalski et al. In this study, the Turkish version of the questionnaire, whose validity and reliability were established by Erdim et al., will be used . The scale evaluates physical activities (PA) performed in the past 7 days and their frequency. Responses are given on a five-point scale, where 5 indicates the highest and 1 the lowest level of physical activity. The total score of the questionnaire is calculated by averaging the scores from 9 questions. A higher score indicates a higher level of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gökşen Kuran Aslan Professor, Phd, Principal Investigator — Istanbul University - Cerrahpasa; Nilay Baş Specialist Physician, Principal Investigator — Istanbul Medicine Faculty
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Faculty of Medicine, Istanbul, Fatih
  - Istanbul Universty Cerrahpaşa, Istanbul, Hadımköy

IPD SHARING:
Plan to Share IPD: No